CLINICAL TRIAL: NCT05208853
Title: An Exploratory Clinical Study Evaluating the Safety and Efficacy of Anti CD30 CAR T Cells Injection (Anti CD30 CAR T Cells) in Patients With CD30+ Relapsed/Refractory Lymphoma
Brief Title: An Exploratory Clinical Study Evaluating the Safety and Efficacy of Anti CD30 CAR T Cells in Patients With CD30+ Relapsed/Refractory Lymphoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Shanghai First Song Therapeutics Co., Ltd (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARM002-CN-2021-01
Record Dates: First submitted 2021-12-24; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Hodgkin Lymphoma; NK/T Cell Lymphoma; Peripheral T Cell Lymphoma, Unspecified; Angioimmunoblastic T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Diffuse Large B Cell Lymphoma; Mediastinal B-Cell Diffuse Large Cell Lymphoma; Gray Zone Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Extranodal NK-T-Cell; Lymphoma, T-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti CD30 CAR T cells (Experimental): Patients receive anti CD30 CAR-T cells on day 0 after lymphodepleting treatment.
  Route of administration: Intravenous injection.
  Lymphodepletion conditioning:
  Lymphodepletion will be conducted several days prior to anti CD30 CAR-T cells infusion.
  Interventions: Biological: Anti CD30 CAR-T Cell Injection

INTERVENTIONS:
Biological: Anti CD30 CAR-T Cell Injection — After enrollment, subjects complete the apheresis, then complete the lymphodepletion, and then receive the dose escalation test: 1.5×10^7 cells，1.5×10^8 cells，5× 10^8 cells.
  Drug: Fludarabine
  Fludarabine is used for lymphodepletion.
  Drug: Cyclophosphamide
  Cyclophosphamide is used for lymphodepletion

SUMMARY:
This is a single-center, open label, single dose study of anti CD30 CAR-T cells injection in treatment of patients with relapsed/refractory CD30+ lymphoma.

DETAILED DESCRIPTION:
This study is a single-center, open-label, single dose study of anti CD30 CAR-T cells injection in treatment of patients with relapsed/refractory CD30+ lymphoma.

This study intends to include CD30-positive patients with relapsed/refractory CD30+ lymphoma, and subjects will receive a single injection of anti CD30 CAR-T cells after screening, Peripheral Blood Mononuclear Cell (PBMC) collection, and lymphodepletion chemotherapy pretreatment. Response assessments for lymphoma subjects will base on 2018 Lugano Classification.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be included in the group:

  1. Understand and sign the informed consent form, and voluntarily participate in clinical study;
  2. 18-70 years old, no gender limit;
  3. Patients with CD30+ lymphoma have received at least 2-line systemic treatment in the past and who have relapsed or are refractory, including but not limited to:

     1. Hodgkins lymphoma;
     2. Mature T-cell lymphoma, including but not limited to non-specific peripheral T cell lymphoma, angioimmunoblastic T-cell lymphoma, NK/T-cell lymphoma, anaplastic large-cell lymphoma;
     3. Diffuse large B-cell lymphoma, including but not limited to mediastinal B-cell lymphoma, gray zone lymphoma;
     4. Other lymphocytic proliferative tumors;
  4. Patients Eastern Cooperative Oncology Group (ECOG) physical status score must be 0 or 1;
  5. Patients with sufficient venous access (for apheresis), and no other contraindications for blood cell separation;
  6. According to the revised version of the efficacy evaluation of malignant lymphoma (2018 lugano standard), Patients should be fluorodeoxyglucose-PET positive and with at least on measurement lesion: long axis of the lesion is ≥ 1.5 cm, or the long axis is 1.0-1.5 cm and short axis ≥1.0cm;
  7. Patients should meet the following laboratory exam requirements during screening, and haven't received cell growth factor (long-acting colony stimulating factor (G-CSF/PEG-CSF) , requires an interval of 2 weeks, except for recombinant erythropoietin) within 7 days before hematological evaluation screening;

     1. The absolute value of neutrophils ≥ 1.0×10^9/L;
     2. Hemoglobin ≥ 90g/L (without red blood cell transfusion within 14 days), hemoglobin in patients with bone marrow involvement ≥ 75g/L;
     3. Platelets in patients without bone marrow involvement≥75×10^9/L, and patients in platelets with bone marrow involvement ≥ 50×10^9/L;
     4. Absolute lymphocyte (ALC) ≥ 0.3×10^9/L;
     5. Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN) (if the bilirubin level rises due to lymphoma invading the liver, allow its total bilirubin ≤ 3 × ULN);
     6. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5×ULN; if AST, ALT elevation is caused by lymphoma invading the liver, allow its AST, ALT ≤ 5×ULN);
     7. Creatinine <1.5 × ULN and endogenous creatinine clearance rate ≥ 60 mL/min;
  8. There is no evidence that the subject has difficulty breathing at rest, and the measured pulse oximetry value when breathing room air is > 90%;
  9. Women of childbearing age must have a negative serum pregnancy test, and they must agree to take effective contraceptive methods at the same time from the signing of the informed consent form to 6 months after the last administration of the study drug.

Exclusion Criteria:

* Patients cannot participate in this study if they meet any of the following conditions:

  1. Patients have a history of allergies to any component in cell therapy products.
  2. Patients received any CAR-T cell product or other genetically modified T cell therapy in the past.
  3. Patients received autologous or allogeneic hematopoietic stem cell transplantation within 3 months.
  4. Patients suffering from other malignant tumors in the past or present (except for skin basal cell carcinoma, breast/cervix carcinoma in situ and other malignant tumors that have not been treated and effectively controlled in the past five years).
  5. Patients who have received continuous systemic steroids (prednisone> 5 mg/day or equivalent doses of other hormones) or other immunosuppressive agents within 14 days before apheresis, except those who have recently or currently used inhaled steroids.
  6. Patients with Hepatitis B (positive hepatitis B virus surface antigen and/or positive hepatitis B core antibody and hepatitis B DNA > 10^3 copies/mL) and Hepatitis C (positive hepatitis C antibody test).
  7. Patients with syphilis, human immunodeficiency virus (HIV) infection (HIV positive).
  8. Patients with hyponatremia and/or hypokalemia, blood sodium < 125 mmol/L and/or blood potassium < 3.5 mmol/L (Except that blood sodium and/or potassium were restored above this level by sodium and/or potassium supplementation before participating in this study).
  9. Patients was known or existing primary or metastatic central nervous system lymphoma, or with any other central nervous system disease (such as seizures, cerebral ischemia/hemorrhage, dementia, etc.).
  10. According to the heart function classification standard of New York Heart Association (NYHA), those with grade III or IV cardiac insufficiency; Cardiac ejection fraction is lower than 50% or lower than the lower limit of the laboratory test value range of the research center, or ECG is significantly abnormal.
  11. Patients with severe respiratory diseases at the time of enrollment (before apheresis), such as interstitial lung disease, active tuberculosis, etc., investigator considered unsuitable for enrollment.
  12. According to the judgment of the investigator, patients with any serious or uncontrollable systemic disease, systemic complications, other serious concurrent diseases (such as hematophilic syndrome, etc.), special tumor conditions may unsuitable for entering this study or affect Protocol compliance, or significant interference with the correct evaluation of the safety, toxicity, and effectiveness of the study drug.
  13. Major surgery has been performed within 4 weeks before apheresis (the definition of major surgery refers to the level 3 and level 4 surgery specified in the "Administrative Measures for the Clinical Application of Medical Technology");Or has not fully recovered from any previous invasive operation.
  14. Patients received systemic chemotherapy within 3 weeks before apheresis, or the toxicity of previous anti-tumor therapy has not recovered ( > CTCAE v5.0 grade 1), except for hair loss and pigmentation.
  15. Patients received Anti-CD30 and other anti-tumor antibody treatments within 4 weeks before apheresis.
  16. Patients received any previous systemic inhibitory/stimulatory immune checkpoint molecular therapy (anti-PD-1/PD-L1 monoclonal antibody), and within 3 half-lives.
  17. Patients have used immunostimulatory or immunosuppressive therapy (such as IFN-α, IFN-β, IL-2, etanercept, infliximab, tacrolimus, cyclosporine or mycophenolic acid) within 28 days before apheresis.
  18. Patients received short-acting targeted therapy (such as tyrosine kinase inhibitors) before apheresis and within 72 hours before infusion.
  19. Those who plan to undergo allogeneic/autologous hematopoietic stem cell transplantation during the study period after the investigators assessment.
  20. Those who have participated in other interventional clinical study before apheresis or within 1 month before administration.
  21. Women who are already pregnant, preparing for pregnant during the study, or breastfeeding.
  22. During the study period, women of childbearing age and men with fertility were unwilling or unable to use reliable contraceptive methods.
  23. Personnel involved in the research plan and implementation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2022-02-10 (Estimated); Primary Completion 2022-02-10 (Estimated); Study Completion 2022-02-10 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | within 4 weeks after infusion
  Maximum Tolerated Dose
AE and SAE | day 0 to month 12
  To evaluate safety of the cell therapy. Adverse event and serious adverse event.

SECONDARY OUTCOMES:
Objective Response Rate, ORR | day 0 to month 12
  Proportion of subjects with complete or partial remission
Disease control rate, DCR | day 0 to month 12
  The percentage of patients with remission and stable disease after treatment in the total evaluable cases.
Duration of remission, DOR | day 0 to month 12
  The time from the first assessment of remission or partial remission of the tumor to the first assessment of disease progression or death from any cause;
Progression-free survival, PFS | day 0 to month 12
  The time from cell reinfusion to the first assessment of tumor progression or death from any cause
Overall survival, OS | day 0 to month 12
  The time from the cell reinfusion to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Huang He, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital, College of medicine, Zhejiang University, Hangzhou, Zhejiang, China